CLINICAL TRIAL: NCT02166879
Title: Undetected Sleep Apnea in the Postanesthesia Acute Care Unit
Brief Title: Undetected Sleep Apnea in the Postanesthesia Acute Care Unit (PACU)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA11-0591
Record Dates: First submitted 2014-06-13; First posted 2014-06-18 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea-Hypopnea Syndrome; Obstructive sleep apnea; OSA; Chart review; Questionnaire; Survey
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS): Chart review from patients undergoing elective surgery.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Participants complete anesthesia questionnaire before elective surgical procedure.
  Other Names: Survey

SUMMARY:
The primary aim is to determine whether patients with suspected OSAHS as predicted by the STOP-BANG questionnaire will have an increased length of stay (LOS) in the postanesthesia acute care unit (PACU) compared with those without suspected OSAHS.

The second aim will be to determine the LOS in patients with known sleep apnea by history. This length of stay will be compared with LOS in patient with an affirmative response to the STOP-BANG questionnaire to determine if prior knowledge of diagnosed sleep apnea will be associated with a lower LOS than in patients with suspected OSA.

The third aim will be to characterize the adverse clinical outcomes (respiratory, cardiovascular, and neurological) associated with suspected OSAHS in patients who respond affirmatively to the STOP-BANG questionnaire and in those patients with known OSA. These data (including number of desaturations, bradypnea, brady- or tachycardia, and use of reversal agents) will be recorded by the PACU nursing staff. Unexpected admissions to the hospital and transfers to the intensive care units will also be measured. These data will help identify the most critical determinants of length of stay.

DETAILED DESCRIPTION:
The study will retrospectively review the anesthetic record, including both the preoperative assessment records and the PACU flow sheets. The study will be conducted in the Anesthesiology Assessment Center. PACU. The STOP-BANG questionnaire is administered as part of the standard of care during the preoperative assessment.

Anesthesia Assessment Center clinics assess approximately 500 patients a week, of which approximately 25% are scheduled for ambulatory surgical procedures in the Mays clinic.

Patients are administered the STOP-BANG questionnaire as part of the standard of care while in the perioperative center. This will be recorded on the Initial Anesthesia Assessment Center Patient Record. This form is filled out by hand by the patients themselves and then scanned into Clinic Station. The neck circumference portion of the Bang questionnaire is assessed and recorded by the medical assistant with the use of a single use disposable paper tape measure. The data are recorded along with basic demographic, historical, and anthropometric data (including BMI) in a preoperative assessment record.

In order to satisfy the first specific aim, length of stay in minutes as determined by the PACU nursing record will be documented. Nurses charting the LOS will not be specifically made aware of the STOP-BANG status of the subjects. Length of stay is charted in the PACU nursing forms electronically in PICIS and relayed to Clinic Station as part of the standard of care for all patients admitted to the PACU.

In order to satisfy the third specific aim, patients enrolled in the study will be monitored for secondary outcomes via chart review of the PACU nursing record and electronic medical record. These outcomes are charted in the PACU nursing forms electronically in PCIS and relayed to Clinic Station as standard of care in all patients in the PACU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients assessed in the Anesthesia Assessment Center who are determined to require same day surgical procedures in the Ambulatory Care Center in the Mays Clinic.
2. Age ≥18

Exclusion Criteria:

1) Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants undergoing elective surgical procedures at UT MD Anderson Cancer Center in Houston, Texas
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2011-09-02 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Length of Stay (LOS) in the Postanesthesia Acute Care Unit (PACU) | 1 day
  Length of stay in minutes as determined by the PACU nursing record documented. A difference in LOS of 15 minutes is considered to be clinically important. A 2-sample t-test used to compare OSAHS risk groups with respect to LOS.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Balachandran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org